CLINICAL TRIAL: NCT00188994
Title: Insulin Cardioplegia Trial for Poor Left Ventricular Function
Brief Title: Insulin Cardioplegia for Poor Left Ventricular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-E089; CIHR Grant No. HSF NA4189
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-07

CONDITIONS: Left Ventricular Dysfunction
Keywords: Myocardial Protection; Myocardial Metabolism; Ventricular Function; Cardiovascular Disease; Cardioplegic Additives
MeSH Terms: conditions — Ventricular Dysfunction, Left; Cardiovascular Diseases

INTERVENTIONS:
Drug: Insulin Cardioplegia

SUMMARY:
The purpose of this investigation is to develop a means to improve the recovery of cardiac metabolism and ventricular function following coronary artery bypass surgery (CABG) in patients with poor preoperative ventricular function (e.g. ejection fraction <40%).

DETAILED DESCRIPTION:
Hypothesis

Insulin added to blood cardioplegia will improve the results of Coronary Artery Bypass Graft by reducing the incidence of low output syndrome (i.e., the requirement for inotropic or balloon pump assistance) in patients with a preoperative ejection fraction <40%.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been referred for isolated coronary bypass surgery.
* LV grade 3 or 4, LVEF <40% by angio, echo, RNA.

Exclusion Criteria:

* Patient is undergoing reoperative surgery (i.e., has had any previous cardiac surgery)
* Surgeon has planned another procedure in addition to coronary bypass surgery (e.g., valve repair, replacement, ascending aorta repair or replacement, left ventricular aneurysm resection, repair of congenital defect, carotid surgery, repair of abdominal aortic aneurysm).
* Patient is scheduled for minimally invasive surgery.
* More recent assessment of LV function with LV grade 1 0r 2, LVEF>40%.
* 5 or 6 days post MI.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800
Dates: Start 1999-08

PRIMARY OUTCOMES:
Low Output Syndrome

SECONDARY OUTCOMES:
Total Troponin I Release

CONTACTS AND LOCATIONS:
Overall Officials: Terrence M. Yau, Principal Investigator — 21st Century Cardiac Surgical Society, Council on Cardiovascular and Thoracic Surgery (American Heart Association), Canadian Cardiovascular Society, Royal College of Physicians and Surgeons, Institute of Medical Sciences (University of Toronto)
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] 1. Yau,TM, Fedak PWM, Weisel RD, Teng C, Ivanov J. Predictors of operative risk for coronary bypass operations in patients with left ventricular dysfunction. J Thorac Cardiovasc Surg 1999; 118:1006-1013. 2. RaoV, Ivanov J, Weisel RD, Ikonomidis JS, Christakis GT, David TE. Predictors of low cardiac output syndrome after coronary artery bypass. J Thorac Cardiovasc Surg 1996; 112:38-51. 3. Yau TM, Weisel RD, Mickle DAG, et al: Optimal delivery of blood cardioplegia. Circulation 1991; 84 (SAuppl II):II-380-388. 4. Yau TM, Weisel RD, Mickle DAG, et al: Alternative techniques of cardioplegia. Circulation 1992; 86(Suppl II):II-377-384. 5. Yau TM, Ikonomidis JS, Weisel RD, et al: Which techniques of cardioplegia prevent ischemia? Ann Thorac Surg 1993; 56:1020-1028. 6. Yau TM, Ikonomiodis JS, Weisel RD, et al: Ventricular function after normothermic versus hypothermic cardioplegia. J Thorac Cardiovasc Surg 1993; 105:883-844. 7. Rao V, Merante F, Weisel RD, Shirai T, Ikonomidis JS, Cohen G, Tumiati LC, Shiono N, Li RK, Mickle DAG, Robinson BH. Insulin stimulates pyruvate dehydrogenase and protects human ventricular cardiomyocytes from simulated ischemia. J Thorac Cardiovasc 1998; 116:485-94. 8. Rao V, Borger MA, Weisel RD, Ivanov J, Christakis GT, Cohen G, Yau TM,. Insulin cardioplegia for elective coronary bypass surgery. J Thorac Cardiovasc Surg 2000; 119: 1176-1184. 9. Yau TM, Mickle DAG, Weisel RD: Myocardial free radical reperfusion injury during cardiac surgery, in Kron IL, Mavroudis C (eds): Frontiers in cardiovascular surgical research: State of Art Reviews: Cardiac Surgery. Hanley & Belfus, 1990; 703-712. 10. Christakis GT, Weisel RD, Fremes SE, Ivanov J, David TE, Goldman BS, Salerno TA and the Cardiovascular Surgeons of the University of Toronto, Coronary Artery bypass grafting in patients with poor ventricular function. J Thorac Cardiovasc Surg 1992; 103:1083-1092.